CLINICAL TRIAL: NCT05362292
Title: Cognitive, Urinary, and Functional Trajectories of Older Women Using Pharmacologic Treatment Strategies for Urgency Incontinence
Brief Title: TReating Incontinence for Underlying Mental and Physical Health
Acronym: TRIUMPH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-35858; 1R01AG075471-01 (NIH)
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence, Urge; Urinary Incontinence; Overactive Bladder; Incontinence, Urge; Incontinence, Urinary; Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence; Urinary Bladder, Overactive | interventions — Tolterodine Tartrate; mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anticholinergic bladder medication plus behavioral self-management education (Active Comparator): Tolterodine tartrate is a muscarinic receptor antagonist designed to treat urgency incontinence, urgency, and frequency associated with overactive bladder. Behavioral self-management education includes written education about timed urination, lifestyle changes, pelvic floor muscle exercises, and urge suppression.
  Interventions: Drug: Tolterodine Tartrate ER
- Beta-3-adrenergic agonist medication plus behavioral self-management education (Active Comparator): Mirabegron, currently sold under the brand name Mybetriq by Astellas Pharma, is a selective beta-3-adrenergic receptor agonist approved for treatment of urgency urinary incontinence, urgency, and frequency associated with overactive bladder. Behavioral self-management education includes written education about timed urination, lifestyle changes, pelvic floor muscle exercises, and urge suppression.
  Interventions: Drug: Mirabegron
- Placebo medication plus behavioral self-management education (Placebo Comparator): Microcrystalline cellulose placebo encapsulated to appear identical to tolterodine and mirabegron medication will be prepared by a compounding pharmacy. Behavioral self-management education includes written education about timed urination, lifestyle changes, pelvic floor muscle exercises, and urge suppression.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolterodine Tartrate ER — Anticholinergic
  Arms: Anticholinergic bladder medication plus behavioral self-management education
Drug: Mirabegron — Beta-3-adrenergic agonist
  Arms: Beta-3-adrenergic agonist medication plus behavioral self-management education
Drug: Placebo — matching placebo pill
  Arms: Placebo medication plus behavioral self-management education

SUMMARY:
The TRIUMPH study is a randomized, double-blinded, 3-arm, parallel-group trial designed to compare the effects of anticholinergic bladder therapy versus a) beta-3-adrenergic agonist bladder therapy and b) no bladder pharmacotherapy on cognitive, urinary, and other aging-related functional outcomes in ambulatory older women with urgency-predominant urinary incontinence and either normal or mildly impaired cognitive function at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older at the time of enrollment
* Female sex at birth, without surgical or hormonal gender re-assignment therapy
* Able to walk to the bathroom and use the toilet without assistance
* Report urinary incontinence starting at least 3 months prior to screening
* Report that at least half of incontinence episodes occur with a sudden or strong sensation of urgency
* Report 2 or more urgency incontinence episodes over a 7-day period
* Willing to provide informed consent and adhere to study procedures throughout the length of the study

Exclusion Criteria:

* Prior clinician diagnosis of dementia, or a Montreal Cognitive Assessment (MOCA) score of 17 or lower on screening cognitive evaluation
* Current use of anticholinergic, beta-3-adrenergic agonist, or other medication designed to improve urgency incontinence symptoms, or use in the past 1 month
* Initiation, discontinuation, or dose change of dementia medications (such as donepezil, galantamine, memantine, rivastigmine) in the past 1 month (but candidates on stable doses are eligible)
* Initiation, discontinuation, or dose change of other drugs with strong anticholinergic effects (based on the Beers List) in the past 1 month (but candidates on stable doses are eligible)
* Initiation, discontinuation, or dose change of other drugs that can affect urinary frequency, including diuretics, in the past 1 month (but candidates on stable doses are eligible)
* Current urinary tract infection (UTI) based on screening urinalysis and culture (but candidates can re-present for re-screening after undergoing treatment for UTI)
* History of allergy or sensitivity to either of the study medications or an ingredient in the placebo or study medication capsule
* Severe hepatic impairment (Child-Pugh score B or greater) or renal impairment (creatinine clearance <30 mL/min) as a contraindication to both study medications
* Current bladder obstruction or urinary retention (defined by symptoms suggesting difficulty emptying the bladder in addition to postvoid residual urine volume greater than 150 cc by portable bladder ultrasound)
* Uncontrolled hypertension (based on measured systolic blood pressure greater than 180 or diastolic blood pressure greater than 110 mmHg) as a contraindication to beta-3-adrenergic therapy
* Self-reported history of gastric retention, uncontrolled narrow angle glaucoma, myasthenia gravis, severe ulcerative colitis, or toxic megacolon as contraindications for anticholinergic bladder therapy
* Use of drugs with adverse interactions with one of the study medications in the past 1 month, including potent CYP3A4 inhibitors, hepatic enzyme metabolism inducers, narrow therapeutic index drugs metabolized by CYP2D6, or intention to start taking one of these medications during the study treatment period
* History of bladder surgery, invasive intra-vesical therapy, or bulk bladder injections in the past 3 months (more remote surgery will not be exclusionary), or intention to undergo one of these procedures in the study treatment period
* Use of other specialized incontinence therapy (electrostimulation, pelvic physiotherapy, formal behavioral therapy overseen by certified practitioners) in the past 3 months (more remote therapy will not be exclusionary), or intention to undergo one of these procedures in the study treatment period
* Inability to sign informed consent or complete questionnaires, interviews, or study testing in English
* Other condition that would prevent the participant from completing study procedures, in the opinion of the investigators (e.g., uncontrolled psychosis)

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 270 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2027-05-02 (Estimated); Study Completion 2027-08-02 (Estimated)

PRIMARY OUTCOMES:
Change in composite cognitive function over 6 months (24 weeks) of treatment, using a composite cognitive score that incorporates normalized data from all domain-specific cognitive tests. | Baseline to 6 months
  The composite cognitive score will be calculated as the average of Z-scores from the following individual cognitive tests: a) Auditory Verbal Learning Test (AVLT); b) Oral Trail Making Test (OTMT) part A; c) OTMT part B; d) Digit Span Test; and e) Digit Symbol Substitution Test (DSST). The normative mean of each cognitive test will be subtracted from each participant's component test score, and this difference will be divided by the standard deviation for the appropriate normative sample. After scores from individual tests are transformed to Z scores as a common metric based on normative data, the average Z score from all available tests will be calculated to provide a composite Z score.

SECONDARY OUTCOMES:
Change in composite cognitive function over 9 months (36 weeks), using a composite cognitive score that incorporates normalized data from all domain-specific cognitive tests. | Baseline to 9 months (3 months after end of treatment)
  The composite cognitive score will be calculated as the average of Z-scores from the following individual cognitive tests: a) Auditory Verbal Learning Test (AVLT); b) Oral Trail Making Test (OTMT) part A; c) OTMT part B; d) Digit Span Test; and e) Digit Symbol Substitution Test (DSST). The normative mean of each cognitive test will be subtracted from each participant's component test score, and this difference will be divided by the standard deviation for the appropriate normative sample. After scores from individual tests are transformed to Z scores as a common metric based on normative data, the average Z score from all available tests will be calculated to provide a composite Z score.
Change in Auditory Verbal Learning Test total learning score assessed over 6 months (24 weeks) of treatment | Baseline to 6 months (end of treatment)
  The Rey Auditory Verbal Learning Test (AVLT), a widely used test of immediate and delayed verbal learning with established norms in older adults and multiple alternate forms. The total learning score is the sum of words learned from trials 1-5.
Change in Auditory Verbal Learning Test total learning score assessed over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  The Rey Auditory Verbal Learning Test (AVLT), a widely used test of immediate and delayed verbal learning with established norms in older adults and multiple alternate forms. The total learning score is the sum of words learned from trials 1-5.
Change Auditory Verbal Learning Test delayed free recall score over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  The Rey Auditory Verbal Learning Test (AVLT), a widely used test of immediate and delayed verbal learning with established norms in older adults and multiple alternate forms. Score range of 0-15.
Change Auditory Verbal Learning Test delayed free recall score over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  The Rey Auditory Verbal Learning Test (AVLT), a widely used test of immediate and delayed verbal learning with established norms in older adults and multiple alternate forms. Score range of 0-15.
Change in Oral Trail Making A score over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  The oral version of the Trail Making Test (OTMT), a timed measure of attention (part A) and executive function (part B) adapted from the written TMT, with established norms for participants across a wide range of ages. Range of 1-150 seconds
Change in Oral Trail Making A score over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  The oral version of the Trail Making Test (OTMT), a timed measure of attention (part A) and executive function (part B) adapted from the written TMT, with established norms for participants across a wide range of ages. Range of 1-150 seconds
Change in Oral Trail Making B score over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  The oral version of the Trail Making Test (OTMT), a timed measure of attention (part A) and executive function (part B) adapted from the written TMT, with established norms for participants across a wide range of ages. Range of 1-300 seconds.
Change in Oral Trail Making B score over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  The oral version of the Trail Making Test (OTMT), a timed measure of attention (part A) and executive function (part B) adapted from the written TMT, with established norms for participants across a wide range of ages. Range of 1-300 seconds.
Change in Digit Span reverse component (total correct trials) over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  The Digit Span Reverse (total correct trials), a subtest of the Wechsler Adult Intelligence and Memory Scales, a test of attention and short-term verbal memory, with reliability across in-person and videoconference platforms. Range of 0-14.
Change in Digit Span reverse component (total correct trials) over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  The Digit Span Reverse (total correct trials), a subtest of the Wechsler Adult Intelligence and Memory Scales, a test of attention and short-term verbal memory, with reliability across in-person and videoconference platforms. Range of 0-14.
Change in Digit Symbol Substitution Test score over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  The Digit Symbol Substitution Test (DSST), a timed, written test assessing incidental memory, visual scanning, and processing speed, in which subjects translate numbers into symbols using a key. Range of 1-133.
Change in Digit Symbol Substitution Test score over 9 months (36 weeks). | Baseline 9 months (3 months after end of treatment)
  The Digit Symbol Substitution Test (DSST), a timed, written test assessing incidental memory, visual scanning, and processing speed, in which subjects translate numbers into symbols using a key. Range of 1-133.
Change in frequency of urgency-type incontinence (episodes/week) over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Frequency and type of incontinence will be assessed using a standardized, 7-day voiding diary.
Change in frequency of urgency-type incontinence (episodes/week) over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Frequency and type of incontinence will be assessed using a standardized, 7-day voiding diary.
Change in frequency of any-type incontinence (episodes/week) over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Frequency and type of incontinence will be assessed using a standardized, 7-day voiding diary.
Change in frequency of any-type incontinence (episodes/week) over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Frequency and type of incontinence will be assessed using a standardized, 7-day voiding diary.
Resolution of urinary incontinence from baseline to 6 months (24 weeks). | Baseline to 6 months (end of treatment)
  Frequency and type of incontinence will be assessed using a standardized, 7-day voiding diary.
Resolution of urinary incontinence from baseline to 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Frequency and type of incontinence will be assessed using a standardized, 7-day voiding diary.
Change in Overactive Bladder Questionnaire Short-Form (OAB-Q SF) Symptom Bother domain score over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Bothersomeness and impact of overactive bladder symptoms (such as urgency, incontinence, and nocturia) will be assessed using the short-form of the OAB-Q, which generates both a Symptom Bother domain and a Health-Related Quality of Life domain score.
Change in Overactive Bladder Questionnaire Short-Form (OAB-Q SF) Symptom Bother domain score over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Bothersomeness and impact of overactive bladder symptoms (such as urgency, incontinence, and nocturia) will be assessed using the short-form of the OAB-Q, which generates both a Symptom Bother domain and a Health-Related Quality of Life domain score.
Change in Overactive Bladder Questionnaire Short-Form (OAB-Q SF) Health-Related Quality of Life domain score over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Bothersomeness and impact of overactive bladder symptoms (such as urgency, incontinence, and nocturia) will be assessed using the short-form of the OAB-Q, which generates both a Symptom Bother domain and a Health-Related Quality of Life domain score.
Change in Overactive Bladder Questionnaire Short-Form (OAB-Q SF) Health-Related Quality of Life domain score over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Bothersomeness and impact of overactive bladder symptoms (such as urgency, incontinence, and nocturia) will be assessed using the short-form of the OAB-Q, which generates both a Symptom Bother domain and a Health-Related Quality of Life domain score.
Change in global sleep quality score over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Perceived sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), an 18-item validated questionnaire designed to assess sleep quality, latency, efficiency, and problems over a one-week period.
Change in global sleep quality score over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Perceived sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), an 18-item validated questionnaire designed to assess sleep quality, latency, efficiency, and problems over a one-week period.
Change in daytime sleepiness score over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS), an 8-item questionnaire assessing the level of general sleepiness during real life situations in order to distinguish excessive daytime sleepiness from normal daytime sleepiness.
Change in daytime sleepiness score over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS), an 8-item questionnaire assessing the level of general sleepiness during real life situations in order to distinguish excessive daytime sleepiness from normal daytime sleepiness.
Change in perceived physical function over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Perceived physical function will be assessed using the PROMIS 10B Adult Physical Function Scale, a 10-item measure that assesses the extent to which daily activities are limited by function of the extremities and central regions.
Change in perceived physical function over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Perceived physical function will be assessed using the PROMIS 10B Adult Physical Function Scale, a 10-item measure that assesses the extent to which daily activities are limited by function of the extremities and central regions.
Change in confidence in maintaining balance over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Confidence in maintaining balance will be assessed using the 15-item Activities Balance Confidence Scale (ABC-S), in which participants self-rate their confidence in keeping balance with performing daily living tasks.
Change in confidence in maintaining balance over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Confidence in maintaining balance will be assessed using the 15-item Activities Balance Confidence Scale (ABC-S), in which participants self-rate their confidence in keeping balance with performing daily living tasks.
Change in overall physical performance over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Physical function will be directly assessed using the Short Physical Performance Battery (SPPB), involving: 1) side-by-side, semi-tandem, and tandem balance tests; 2) a 4-meter walk test; and 3) 5 chair stands, in which participants will be asked to stand up repeatedly from a standard chair to a full extended standing position.
Change in overall physical performance over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Physical function will be directly assessed using the Short Physical Performance Battery (SPPB), involving: 1) side-by-side, semi-tandem, and tandem balance tests; 2) a 4-meter walk test; and 3) 5 chair stands, in which participants will be asked to stand up repeatedly from a standard chair to a full extended standing position.
Change in static balance over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Static balance will additionally be assessed by asking participants to attempt to assume a one-legged stand for 30 seconds.
Change in static balance from over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Static balance will additionally be assessed by asking participants to attempt to assume a one-legged stand for 30 seconds.
Change in lower extremity strength measured by chair stand testing over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Physical strength will be assessed 30-second chair stand, by asking participants to stand up as many times as possible within 30 seconds, with higher number indicating more strength or power.
Change in lower extremity strength measured by chair stand testing over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Physical strength will be assessed 30-second chair stand, by asking participants to stand up as many times as possible within 30 seconds, with higher number indicating more strength or power.
Change in depression symptoms over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Depression symptoms will be assessed using the 15-item short form of the Geriatric Depression Scale-15 (GDS-15), which assesses symptoms of depression over a 1-week period.
Change in depression symptoms over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Depression symptoms will be assessed using the 15-item short form of the Geriatric Depression Scale-15 (GDS-15), which assesses symptoms of depression over a 1-week period.
Change in anxiety symptoms over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Anxiety symptoms will be assessing using the Generalized Anxiety Disorder-7 (GAD7), 7-item short form, questionnaire to assess severity of anxiety symptoms over a 2-week period.
Change in anxiety symptoms over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Anxiety symptoms will be assessing using the Generalized Anxiety Disorder-7 (GAD7), 7-item short form, questionnaire to assess severity of anxiety symptoms over a 2-week period.
Change in constipation symptoms over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Symptoms of constipation as a possible side effect of anticholinergic therapy will be assessed by the 9-item PROMIS Constipation scale of the PROMIS Gastrointestinal Symptoms-Constipation Scale.
Change in constipation symptoms over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Symptoms of constipation as a possible side effect of anticholinergic therapy will be assessed by the 9-item PROMIS Constipation scale of the PROMIS Gastrointestinal Symptoms-Constipation Scale.
Change in bowel incontinence symptoms over 6 months (24 weeks) of treatment. | Baseline to 6 months (end of treatment)
  Bowel incontinence as a syndrome that frequently overlaps with urinary incontinence will be assessed using the 4-item PROMIS Bowel Incontinence scale.
Change in bowel incontinence symptoms over 9 months (36 weeks). | Baseline to 9 months (3 months after end of treatment)
  Bowel incontinence as a syndrome that frequently overlaps with urinary incontinence will be assessed using the 4-item PROMIS Bowel Incontinence scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MD, MAS, MPhil, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
The investigative team will make publicly available de-identified individual participant data that underlie the results reported in the publication. This will include data about the baseline characteristics of enrolled participants and any primary or secondary trial outcomes presented in the publication. To gain access, data requestors will be asked to sign a data access agreement.
Supporting Information: ICF
Time Frame: Starting no later than 6 months following publication of the main trial results (including on-line publication), the investigative team will make publicly available de-identified individual participant data that underlie the results reported in the publication. This will include data about the baseline characteristics of the study participants and any primary or secondary trial outcomes presented in the publication.

REFERENCES:
- [Derived] Huang AJ, Walter LC, Yaffe K, Vittinghoff E, Kornblith E, Schembri M, Chang A, Subak LL. TReating Incontinence for Underlying Mental and Physical Health (TRIUMPH): a study protocol for a multicenter, double-blinded, randomized, 3-arm trial to evaluate the multisystem effects of pharmacologic treatment strategies for urgency-predominant urinary incontinence in ambulatory older women. Trials. 2023 Apr 21;24(1):287. doi: 10.1186/s13063-023-07279-z. PMID 37085880